CLINICAL TRIAL: NCT02243033
Title: A Phase II Study to Evaluate Outpatient Magnetic Resonance Image-guided Laser Focal Therapy for Prostate Cancer, a 20-year Survival Study
Brief Title: Phase II Laser Focal Therapy of Prostate Cancer
Acronym: LITT or FLA
Status: Active, not recruiting | Type: Observational
Sponsor: HALO Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: DMI-Laser-001; WIRB Pr. No.: 20140945 (Other: Western Institutional Review Board)
Record Dates: First submitted 2014-09-09; First posted 2014-09-17 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Focal therapy; Laser therapy; Transrectal; MRI-guided
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Visualase: MR-guided laser focal therapy
  Interventions: Device: MR-guided laser focal therapy

INTERVENTIONS:
Device: MR-guided laser focal therapy — Placement of laser applicator under MRI guidance and real-time MR thermal imaging of tissue necrosis.
  Other Names: Visualase; Tranberg

SUMMARY:
Target recruitment: 1000 subjects. The purpose of this research study is to continue to investigate the safety and effectiveness of using MR (magnetic resonance) guided laser focal therapy for prostate cancer and to evaluate oncologic control over 20 years. We hypothesize that laser focal therapy can be used to achieve oncologic control in carefully selected patients.

MR uses large magnets to produce pictures of areas/organs inside the body. The laser uses light to heat a target area to try to destroy cancerous cells.

The laser system that will be used is called the Visualase® Thermal Therapy System. This system has been used for the treatment of brain, bone (spine), thyroid, and liver cancers. However; this study is the first time this system has been studied for use in the treatment of prostate cancer with a trans-rectal approach.

MR-guided biopsies and laser applicator placement will be performed using the Invivo DynaTRIM trans-rectal biopsy guidance system. This system is cleared (approved) by the U.S. Food and Drug Administration (FDA) for such uses.

DETAILED DESCRIPTION:
Laser-induced interstitial thermal therapy (LITT) is a novel form of controlled, targeted thermal ablation that may offer measurable advantages over other ablative therapies for focal prostate therapy. Because LITT is magnetic resonance (MR) compatible, it enables an imaging advantage over other surgical or ablation techniques that utilize transrectal ultrasound to target and monitor treatment. MR imaging provides excellent soft-tissue contrast and three-dimensional (3D) anatomical imaging in any arbitrary plane, which can help to improve treatment planning and targeting. Additionally, MR-based temperature monitoring allows real-time feedback during MRI-guided thermal therapy as both deposition of light energy and MR signal acquisition can be performed simultaneously without degradation in the MR signal. Also, being in the MR diagnostic environment allows use of post- treatment imaging to verify tissue damage. Because MR images clearly depict the prostate anatomy and the surrounding critical structures, MR imaging has been incorporated into planning for external- beam radiotherapy, brachytherapy, and other treatments of the prostate. In addition to these basic features, Multiparametric prostate MRI (mpMRI) may be used to identify regions of disease in the prostate and better target therapy.

In this study, the investigators propose to evaluate the efficacy of a novel, FDA-approved thermal therapy and feedback system (Visualase® Thermal Therapy System) for the treatment of biopsy confirmed and MR-imageable prostate lesions. This system has been used in humans for the treatment of brain, bone (spine), thyroid, and liver cancers. Early feasibility studies for prostate cancer used a transperineal approach; however it is now being evaluated for the primary treatment of prostate cancer using a transrectal approach. This system allows delivery of laser energy while the patient is simultaneously being imaged by an MRI unit. The system's real-time MR thermal imaging (MRTI) provides information on the thermal dose delivered to the target, resulting in a more precise and controlled delivery which has previously not been possible with other ablative therapies. The investigators hypothesize the system can be integrated into a practical and feasible outpatient treatment paradigm for focal treatment of localized prostate cancer and allow patients to avoid the complications associated with radical whole-gland therapy.

ELIGIBILITY:
Inclusion Criteria:

Treatment Naïve patients:

* Male, 45 years of age or older.
* Diagnosis of prostate adenocarcinoma.
* Clinical stage T1c or T2a.
* Gleason score of 7 (3+4 or 4+3) or less.
* Three or fewer biopsy cores with prostate cancer.
* PSA density not exceeding 0.375.
* One, two, or three tumor suspicious regions identified on multiparametric MRI.
* Negative radiographic indication of extra-capsular extent.
* Karnofsky performance status of at least 70.
* Estimated survival of 5 years or greater, as determined by treating physician.
* Tolerance for anesthesia/sedation.
* Ability to give informed consent.
* At least 6 weeks since any previous prostate biopsy.
* MR-guided biopsy confirmation of one or more MRI-visible prostate lesion(s) with Gleason score of 7 (3+4 or 4+3) or less.

Salvage candidates will be accepted upon physician referral.

Exclusion Criteria:

* Presence of any condition (e.g., metal implant, shrapnel) not compatible with MRI.
* Severe lower urinary tract symptoms as measured by an International Prostate Symptom Score (IPSS) of 20 or greater
* History of other primary non-skin malignancy within previous three years.
* Diabetes
* Smoker

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-05; Primary Completion 2036-05 (Estimated); Study Completion 2036-11 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events | 1 yr. post treatment
  Number of subjects reporting serious adverse events.

SECONDARY OUTCOMES:
Efficacy of treatment | 1 yr. post treatment
  MR-guided biopsy results of treated area and PSA.

OTHER OUTCOMES:
Time to biochemical recurrence | Up to 20 years
  PSA measurement
Time to metastasis | Up to 20 years
  Imaging utilizing PET/CT or other modality
Cause of death | Up to 20 years
  Death certificate or report from partner/spouse/primary care physician

CONTACTS AND LOCATIONS:
Overall Officials: John F. Feller, MD, Principal Investigator — HALO Diagnostics; Bernadette M. Greenwood, MSc, Study Director — HALO Diagnostics
Locations (1):
- Desert Medical Imaging, Indian Wells, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Bi-annaually at the meetings of the International Laser Network until study closure.
Access Criteria: Scientists and physicians studying or performing laser focal therapy.

REFERENCES:
- [Background] Greenwood, B. et al.: Transrectal interventional MRI: initial prostate biopsy experience. SPIE Proceedings, 2010.
- [Background] Hakimi AA, Feder M, Ghavamian R. Minimally invasive approaches to prostate cancer: a review of the current literature. Urol J. 2007 Summer;4(3):130-7. PMID 17987573
- [Background] Menon M, Tewari A, Peabody JO, Shrivastava A, Kaul S, Bhandari A, Hemal AK. Vattikuti Institute prostatectomy, a technique of robotic radical prostatectomy for management of localized carcinoma of the prostate: experience of over 1100 cases. Urol Clin North Am. 2004 Nov;31(4):701-17. doi: 10.1016/j.ucl.2004.06.011. PMID 15474597
- [Background] Valerio M, Emberton M, Ahmed HU. Focal therapy will become a standard option for selected men with localized prostate cancer. J Clin Oncol. 2014 Nov 10;32(32):3680-1. doi: 10.1200/JCO.2014.56.7792. Epub 2014 Aug 18. No abstract available. PMID 25135989
- See also: HALODx — http://www.halodx.com